CLINICAL TRIAL: NCT04037839
Title: High Flow Nasal Cannula Therapy in the Paediatric Home Setting
Brief Title: Nasal High Flow Therapy in the Paediatric Home Setting
Acronym: HFNC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Patrick Stafler, Senior Pulmonologist, Rabin Medical Center
Other Study IDs: Vapotherm
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Disease; Lung Diseases
MeSH Terms: conditions — Respiration Disorders; Lung Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Medical records of children aged 0-18 years who were prescribed a HFNC device at Schneider Children's between 2014-2018 for use in the home setting will be reviewed retrospectively. As part of the telephone consent process, parents will be offered to "opt out" at the beginning of the interview.

SUMMARY:
High flow nasal cannula (HFNC) therapy is non-invasive respiratory support designed to deliver a high flow of heated humidified air, with or without entrained oxygen, via specifically designed nasal prongs. Initially developed for preterm infants, the application of the technology is rapidly spreading to include pediatric patients with various indications, including bronchiolitis, obstructive sleep apnea (OSA), tracheomalacia, asthma, post- extubation support, and even adult hypoxemic respiratory failure.

Since it appears to be better tolerated than traditional modes of non-invasive ventilation, such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), it is increasingly used outside the intensive care setting, despite limited evidence of its safety and efficacy. In Israel, HFNC is approved for home support of children requiring non-invasive respiratory support on the recommendation of a paediatric pulmonologist or intensivist, provided that CPAP and BiPAP have been trialed and deemed not tolerated by the patient.

At Schneider Childrens' Medical Center of Israel (SCMI), a tertiary paediatric hospital, therapy is commenced during a brief inpatient stay, at a period of clinical stability. Parents are trained in the use of the device and flow rate is titrated to clinical response.

The investigators aim to describe the safety, indications, parameters of utilization, length of treatment, clinical outcomes and parental satisfaction of HFNC in the paediatric home setting.

DETAILED DESCRIPTION:
High flow nasal cannula (HFNC) therapy is non-invasive respiratory support designed to deliver a high flow of heated humidified air, with or without entrained oxygen, via specifically designed nasal prongs. Its physiological benefits include flow-dependent positive airway pressure, alveolar recruitment and washout of carbon dioxide from the upper airway. The reduction of esophageal pressure changes during respiration, compared with standard non-occlusive oxygen facemask, indicates its capacity to ease inspiratory effort.

Initially developed for preterm infants, the application of this technology is rapidly spreading to include pediatric patients with various indications, including bronchiolitis, obstructive sleep apnea (OSA), tracheomalacia, asthma, post-extubation support, and even adult hypoxemic respiratory failure.

Since it appears to be better tolerated than traditional modes of non-invasive ventilation, such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), it is increasingly used outside the intensive care setting, despite limited evidence of its safety and efficacy.

In Israel, HFNC is approved for home support of children requiring non-invasive respiratory support on the recommendation of a paediatric pulmonologist or intensivist, provided that CPAP and BiPAP have been trialed and deemed not tolerated by the patient. At Schneider Childrens' Medical Center of Israel (SCMI), a tertiary paediatric hospital, therapy is commenced during a brief inpatient stay, at a period of clinical stability. Parents are trained in the use of the device and flow rate is titrated to clinical response.

The investigators aim to describe the safety, indications, parameters of utilization, length of treatment, clinical outcomes and parental satisfaction of HFNC in the paediatric home setting.

Medical records of children aged 0-18 years who were prescribed a HFNC device at Schneider Children's between 2014-2018 for use in the home setting will be reviewed retrospectively. Demographic and clinical data will be collected. This will be supplemented by a standardized telephone questionnaire. Verbal consent will be obtained from one of the parents, and documented. As part of the telephone consent process, parents will be offered to "opt out" at the beginning of the interview.

ELIGIBILITY:
Inclusion Criteria:

1. Any child who received HFNC
2. Previously trialed CPAP and BiPaP and deemed not tolerated by patient.

Exclusion Criteria:

N/A

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Preterm infants and pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in cumulative days of hospital admission | 6 months before compared to 6 months after starting high flow nasal cannula treatment
  For all participants, 2 periods will be compared in terms of days of hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stafler, Principal Investigator — Schneider Children's
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No